CLINICAL TRIAL: NCT02386878
Title: The Effectiveness of Two Promising Interventions for Reducing HIV Risk and Improving the Wellbeing of Orphaned and Vulnerable Adolescents in the Eastern Cape of South Africa
Brief Title: HIV/AIDS Orphaned and Vulnerable Children Public Health Evaluation
Acronym: PHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University School of Social Work (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Tonya Renee Thurman, Principle Investigator, Tulane University School of Social Work
Organization: Tulane University (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: PHE# ZA.09.0257
Record Dates: First submitted 2015-03-06; First posted 2015-03-12 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Adolescent Behavior; Risk Reduction Behavior; Stress, Psychological
Keywords: Orphans and vulnerable children (OVC); Program Evaluation; HIV Prevention; Psychosocial Wellbeing; Adolescents
MeSH Terms: conditions — Adolescent Behavior; Risk Reduction Behavior; Stress, Psychological | interventions — Interpersonal Psychotherapy; Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Interpersonal Psychotherapy for Groups (IPTG) (Experimental): The intervention consists of 16 weekly 60 to 90 minute psychotherapy sessions, implemented once a week by a trained lay facilitator.
  Interventions: Behavioral: Interpersonal Psychotherapy for Groups (IPTG)
- Vhutshilo 2 (Experimental): The intervention consists of 13 group sessions, implemented once a week by a trained lay facilitator.
  Interventions: Behavioral: Vhutshilo 2
- IPTG and Vhutshilo (Experimental): Participants receive the IPTG intervention first, followed by Vhutshilo 2.
  Interventions: Behavioral: Interpersonal Psychotherapy for Groups (IPTG); Behavioral: Vhutshilo 2
- No Intervention (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy for Groups (IPTG) — Interpersonal psychotherapy is a theory- and evidence-based treatment approach for depression developed by clinicians. World Vision has helped to pioneer the use of this model in sub-Saharan Africa including adapting the model for use with OVC within South Africa. Sessions are designed to provide participants with opportunities to learn and practice interpersonal skills for solving problems that bring about depression, and to facilitate the provision of emotional support between members of the group. Groups are implemented by a trained adult facilitator from the community who helps participants to identify people who are important in their lives, understand links between their psychological state and current problems, and practice new ways of problem-solving.
  Arms: IPTG and Vhutshilo; Interpersonal Psychotherapy for Groups (IPTG)
Behavioral: Vhutshilo 2 — The Vhutshilo 2 model was developed in 2008 by the Centre for the Support of Peer Education (CSPE), a branch of the South African non-profit organization Health and Education Training and Technical Assistance Services. The Vhutshilo program was designed specifically for adolescent OVC in South Africa, and attends to risk factors and pathways considered particularly relevant for this population. Topics include finding and giving emotional support; dealing with grief and loss; alcohol and substance abuse; crime and sexual violence; HIV/AIDS; healthy and safe sexual relationships; and transactional sex. In addition to its knowledge component, the program places heavy emphasis on building relevant skills and efficacy.
  Arms: IPTG and Vhutshilo; Vhutshilo 2

SUMMARY:
The PHE study is a two-year longitudinal study evaluating two interventions for reducing depression and HIV risk behaviors among highly vulnerable adolescents in the Eastern Cape of South Africa. Research suggests that children affected by AIDS are at heightened risk of HIV infection relative to their peers; however, evidence on how best to address HIV prevention and psychological health among this population is lacking. This study examines the efficacy of both a psychological and behavioral intervention, alone and in combination, on related outcomes among vulnerable youth age 14-17. A mixed methods approach is applied, including a community-randomized controlled trial with a factorial design, a cost-effectiveness analysis, and a qualitative component. At baseline data collection in January 2012, more than 1000 adolescents and their caregivers were interviewed; these participants were invited to take part in two more survey rounds designed to examine both the immediate and long term effects of the interventions. Support for this research was provided by USAID under Grant No. GHH-I-00-007-00069-00.

DETAILED DESCRIPTION:
The study will apply a mixed-methods approach involving two primary components: 1) an impact evaluation using a community-randomized controlled trial (CRCT); and 2) a detailed analysis of intervention costs, linked to the impact evaluation to determine the cost-effectiveness of these interventions.

For the CRCT, sixty World Vision drop-in centers which deliver standard care were randomly assigned to one of four study conditions: IPTG, Vhutshilo, IPTG+Vhutshilo, and control. Approximately 1600 adolescent OVC aged 14-17 years (current beneficiaries at the drop-in centers) and their caregivers were eligible to participate in the study at baseline.

Participants were visited three times including the baseline survey. Follow-up data collection was conducted in two rounds. The first round took place 8 months after the baseline survey and immediately following intervention exposure. A second follow-up round took place a year later, allowing assessment of both the immediate and longer-term impact of the interventions.

Participants were interviewed at home in Xhosa or Sesotho. Caregivers in the sample completed face-to-face interviews with trained interviewers, while adolescents complete surveys used a mix of face-to-face interviewing and audio computer-assisted self-interview technology (ACASI).

ELIGIBILITY:
Inclusion Criteria:

* Aged 14-17 years old as of January 1, 2012;
* Enrolled in a selected World Vision site;
* Willing and able to assent to study participation; and
* Consent given by the parent or guardian for the adolescent to participate in the study.

Exclusion Criteria:

* Are not able to give informed assent due to known or recognizable cognitive or psychiatric impairment.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2302 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in Sexual Risk Behavior | Baseline, 0 months post-intervention, 12 months post intervention
  Adolescent self-report of key sexual behaviors including age at sexual debut; the number of sexual partners; and whether condoms were used consistently in the last 6 months.
Change in Depressive Symptoms | Baseline, 0 months post-intervention, 12 months post intervention
  Adolescent self-report of the 20-item Center for Epidemiologic Studies Depression Scale for children (CES-DC). The response options used for the CES-DC are on a 4-point scale (not at all; a little; some; a lot).

SECONDARY OUTCOMES:
Change in HIV knowledge | Baseline, 0 months post-intervention, 12 months post intervention
  Adolescent self-report of basic HIV knowledge: 9 items were used to measure general HIV transmission, testing and treatment knowledge. Respondents were asked to agree or disagree with each item. They could also respond with 'don't know'. The first item (testing for HIV) came from the UNDP/UNFPA/WHO/World Bank Special Programme of Research, Development and Research Training in Human Reproduction (HRP)'s Asking Young People about Sexual And Reproductive Health (HIV testing). Four items, including transmission by mosquitoes, sharing food, witchcraft, and healthy-looking person with HIV, were from the South African Demographic and Health Survey. Two items were pulled from a previous evaluation of Vhutshilo 2 in South Africa (perinatal transmission, sex with a virgin). Two questions were self-generated to gather knowledge of drug treatment availability and exact location of VCT site.
Change in Condom Knowledge and Attitudes | Baseline, 0 months post-intervention, 12 months post intervention
  Adolescent self-report of three items assessing condom knowledge and three items assessing condom attitudes. Respondents indicated agree, disagree or don't know for each item. The South Africa DHS provided two condom knowledge items, whether the male condom provides protection from HIV and whether condoms can be washed and reused. The third knowledge item, whether condoms can be used with Vaseline, came from the South Africa and Tanzania project (SATZ) questionnaire. The SATZ questionnaire also provided one of the three items to measure attitudes toward condom use, which is particularly useful for its gendered perspective; the question asks whether it is okay for a girl to suggest condom use to a sexual partner. The other two items assessing attitudes, including embarrassment and trust, are from the Stepping Stone Study men's questionnaire.
Change in Peer Norms | Baseline, 0 months post-intervention, 12 months post intervention
  Adolescent self-report of three self-generated items with the stem "Many friends your age are…" These items were used to assess peer norms regarding sexual activity, condom use and peer expectations. Respondents indicated agree, disagree or don't know for each item.
Change in Self-Efficacy | Baseline, 0 months post-intervention, 12 months post intervention
  Adolescent self-report of six items adapted from the SATZ Women's Questionnaire. Using a 4-point Likert scale (very low to very high), they ask "what are the chance you would be able…" regarding condom use (3 items) and refusal to have sex (3 items).
Change in Social Support | Baseline, 0 months post-intervention, 12 months post intervention
  Evidence suggests that social support is a mediator of depression symptom severity. Four items were used to assess social support (friends and people in your life) using the 4-point scale from the CES-DC (not at all; a little, some, a lot). Adolescent self-report of four items adapted from the Interpersonal Support Evaluation List (ISEL).
Change in Future Expectations | Baseline, 0 months post-intervention, 12 months post intervention
  Adolescent self-report of six items assessing future expectations. Participants were asked "what are the chances that you will…" fulfill each of six items (marriage, children, secondary school, long life, manage difficulties, job) on a 4-point Likert scale (very low to very high). The items were based on two scales; one is a self-generated scale used in a previous study of OVC in South Africa by the authors and the other is an adapted subscale of the Social and Health Assessment (SAHA) previously used among South African adolescents.
Change in Alcohol Use | Baseline, 0 months post-intervention, 12 months post intervention
  Adolescent self-report of two items. The SA DHS provided an item to assess alcohol use ever, while frequency of alcohol use (last 6 months) was measured using an item from Transitions study.
Change in VCT | Baseline, 0 months post-intervention, 12 months post intervention
  Adolescent self report of two items measuring whether the participant has received an HIV test (ever and last six months) were adapted from Transitions and self-generated respectively.
Change in STI | Baseline, 0 months post-intervention, 12 months post intervention
  Adolescent self report on of sores on or abnormal discharge from their penis/vagina. Symptoms of an STI was measured with one question modified from Transitions.

OTHER OUTCOMES:
Demographic Information | Baseline, 0 months post-intervention, 12 months post intervention
  Adolescent self-report of age. Caregiver report of age, marriage status, education level, and relationship to adolescent. Interviewer observation of race and gender
Adolescent Education | Baseline, 0 months post-intervention, 12 months post intervention
  Current attendance and grade level were measured using items modified from the SA DHS. A self-generated question was used to measure school absenteeism.
Adolescent Health | Baseline, 0 months post-intervention, 12 months post intervention
  Adolescent self-report of five items measuring health. Self-rated health was measured using question G1.2 of the World Health Organization's Quality of Life-100 instrument (WHOQOL-100). Morbidity, including illnesses common to South Africa was measured using an abbreviated scale from The Young Carers Project South Africa survey.
Traumatic Events | Baseline, 0 months post-intervention, 12 months post intervention
  Adolescent self-report of personal experience with HIV (experience and relationship to someone infected with or deceased from HIV/AIDS); emotional maltreatment in the home; and bullying/social isolation (how often other kids make fun of the youth). Caregiver report of adolescent's contact with parents; parental illness and death (including AIDS-specific verbal autopsy); and household illness and deaths burden in last year (including economic impact)
Caregiver Health | Baseline, 0 months post-intervention, 12 months post intervention
  Self-rated health and a modified AIDS-specific verbal autopsy
Caregiver Psychological Health | Baseline, 0 months post-intervention, 12 months post intervention
  Caregiver self-report of depressive symptomology using the the Center for Epidemiological Studies Depression 10 item scale (CESD-10)
Caregiver Social Relationships | Baseline, 0 months post-intervention, 12 months post intervention
  Caregiver self-report of items measuring Social support; Caregiving burden for orphans and for ill household members; Perceived community stigma; and monitoring of adolescent behavior.
Caregiver HIV Knowledge, Attitudes and Communication | Baseline, 0 months post-intervention, 12 months post intervention
  Caregiver self-report of items measuring HIV transmission methods; Rejection of major HIV misconceptions; Attitudes towards sex and reproductive health education; and communication with adolescent pertaining to sexuality and HIv

CONTACTS AND LOCATIONS:
Overall Officials: Tonya R Thurman, MPH PhD, Principal Investigator — Tulane University School of Social Work

REFERENCES:
- [Derived] Thurman TR, Nice J, Taylor TM, Luckett B. Mitigating depression among orphaned and vulnerable adolescents: a randomized controlled trial of interpersonal psychotherapy for groups in South Africa. Child Adolesc Ment Health. 2017 Nov;22(4):224-231. doi: 10.1111/camh.12241. Epub 2017 Sep 26. PMID 32680417